CLINICAL TRIAL: NCT04258007
Title: Recovery Profile of Sugammadex Versus Neostigmine in Pediatric Patients Undergoing Cardiac Catheterization: a Randomized Double-blind Study
Brief Title: Sugammadex Versus Neostigmine in Pediatric Less Than Two Years Undergoing Cardiac Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS.19.08.759
Record Dates: First submitted 2020-01-28; First posted 2020-02-06 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Cardiac Catheterization
MeSH Terms: interventions — Neostigmine; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double blind (Participant, Care Provider)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reversal Neostigmine (Placebo Comparator): Patients undergoing cardiac catheterization will receive a combination of 0.02 mg/ kg atropine and 0.04 mg/ kg neostigmine following observing the second response on stimulating the ulnar nerve on the TOF watch
  Interventions: Drug: Reversal Neostigmine
- Reversal Sugammadex (Active Comparator): Patients undergoing cardiac catheterization will receive sugammadex 4 mg/ kg when the T2 is observed on the TOF watch
  Interventions: Drug: Reversal Sugammadex

INTERVENTIONS:
Drug: Reversal Neostigmine — Patients will receive 0.02 mg/ kg atropine and 0.04 mg/ kg neostigmine following observing the second response on stimulating the ulnar nerve on the TOF watch
  Other Names: PROSTIGMIN®
  Arms: Reversal Neostigmine
Drug: Reversal Sugammadex — Interventional Arm Patients undergoing cardiac catheterization will receive sugammadex 4 mg/ kg when the T2 is observed on the TOF watch
  Other Names: BRIDION®
  Arms: Reversal Sugammadex

SUMMARY:
This study hypothesizes that Sugammadex may has more appropriate recovery profile than neostigmine in pediatric cardiac patients undergoing cardiac catheterization. In pediatric cardiac patients, clear and rapid recovery (fast-tracking) is required to maintain hemodynamic within the normal physiological values which may be saved by sugammadex

DETAILED DESCRIPTION:
There are numerous advantages of early tracheal extubation otherwise known as fast-tracking following anesthesia for congenital heart disease (CHD)

Early tracheal extubation not only eliminates the potential morbidity related to an endotracheal tube and mechanical ventilation such as atelectasis, accumulation of secretions, nosocomial infections, and the potential for airway trauma, it also limits the need for sedation and the antecedent adverse effects including respiratory and hemodynamic depression, tolerance, withdrawal, and delirium. Most importantly, the shift from positive pressure to spontaneous ventilation augments cardiovascular function and improves preload. Reversal of neuromuscular blockade is a fundamental aspect of emergence from general anesthesia. Historically, the only option to actively reverse blockade will be to administer anticholinesterase inhibitors, which are unable to reverse deep neuromuscular blockade. They are also associated with a variety of cholinergic side effects, including bradycardia, nausea, and increased secretions, which require concomitant administration of an anticholinergic agent, with its own adverse effects. Sugammadex is a newer, selective relaxant binding agent

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status (ASA) I-III

Exclusion Criteria:

* Legal guardian refusal.
* Any patients with known drug hypersensitivity.
* Kidney failure.
* Liver failure.
* Diseases affecting the neuromuscular junction.
* A history of malignant hyperthermia

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Reversal efficacy | 90 minutes after endotracheal extubation
  Mean time in minutes from start of sugammadex or neostigmine administration to recovery of T4/T1 ratio to 0.9 was assessed by applying repetitive train of four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. Nerve stimulation continued until the ratio of the magnitude of the fourth twitch (T4) to first twitch (T1) reached at least 0.9

SECONDARY OUTCOMES:
Heart rate | assessed basal, after induction, every 15 min during operation ,.just before reversal, and at 1,2,5,7,10,15 minutes after reversal
Mean arterial blood pressure | basal, after induction, every 15 min during operation ,.just before reversal, and at 1,2,5,7,10,15 minutes after reversal
Diastolic arterial blood pressure | basal, after induction, every 15 min during operation ,.just before reversal, and at 1,2,5,7,10,15 minutes after reversal
Peripheral oxygen saturation | basal, after induction, every 15 min during operation , just before reversal, at 1,2,5,7,10,15 minutes after reversal
vomiting | for 24 hour after sugammadex or neostigmine administration
  patients monitored for incidence and rate of vomiting by clinical observation in PACU for 24 hours after sugammadex or neostigmine administration .
Anaphylaxis | for 24 hour after sugammadex or neostigmine administration
  patients monitored after sugammadex or neostigmine administration for 24 hours postoperative for The National Institute of Allergy and Infectious Diseases (NIAID) and the Food Allergy and Anaphylaxis
  Network (FAAN) proposed clinical criteria for diagnosing anaphylaxis . Depending on the severity of the reaction, four grades of immediate clinical manifestations are described:
  Grade 1, Cutaneous signs only; Grade 2, Measurable but not life-threatening symptoms and cutaneous signs,hypotension, tachycardia, and respiratory disturbances, such as cough and difficulty in lung inflation; Grade 3, Life-threatening symptoms: collapse, tachycardia or bradycardia, arrhythmias, bronchospasm; Grade 4, Cardiac and/or respiratory arrest
blood glucose | preoperative, 15 minutes before reversal and 30 minutes after reversal
  blood glucose in (mg/dL) measured using a GLUCOMETER with strip
prothrombin time | intraoperative and for 60 minutes after sugammadex or neostigmine administration
  PT in seconds measured Just before reversal and 60 min after reversal administration.
activated prothromboplastin time | intraoperative and for 60 minutes after sugammadex or neostigmine administration
  APTT in seconds measured Just before reversal and 60 min after reversal administration.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif A Mousa, MD, Study Chair — Professor of Anaesthesia and Surgical Intensive Care; Amgad A Zaghloul, MD, Study Director — Associate Professor of Anaesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Following publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: forever
Access Criteria: ahmed.refaat.rezk@gmail.com